CLINICAL TRIAL: NCT00498888
Title: Is the a Difference Between Rehabilitation Treatment, Pelvic Floor Muscle Training, Bladder Training and Anticholinergic Drug Treatment in UUI in the Long Term: A Study of Impairment, Quality of Life, and Cost Effectiveness
Brief Title: The Long Term Outcomes of Rehabilitation and Drug Treatment for in Urgency Urinary Incontinence
Acronym: UUI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Hospital Systems (Other)
Responsible Party: Principal Investigator, rachel kafri, Maccabi Healthcare Services, Assuta Hospital Systems
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2007030
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Urge Urinary Incontinence
Keywords: urge urinary incontinence; rehabilitation; anticholinergic
MeSH Terms: conditions — Urinary Incontinence, Urge | interventions — Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Active Comparator): Women were prescribed a 3 month supply of Tolterodine SR 4 mg (Detrusitol SR 4 mg, Pfizer Pharmaceuticals Israel LTD) . After the randomization she needs to get the first prescription from her doctor, and followed this protocol every three weeks. Her doctor how already knows this research were explained how to take the drug. After finished this protocol she get the money she pay after sending the receipts and the empty boxes.
  Interventions: Procedure: tolterodine
- 2 (Active Comparator): The Bladder training protocol aims o to increase the time interval between voids, either by a mandatory or self-adjustable schedule, so that incontinence is ultimately avoided and continence regained. It is generally comprised of three components: 1) patient education that includes information about bladder and how continence is usually maintained, 2) scheduled voiding- a 'timetable for voiding' which may fixed or flexible to suit the participant's rate of increase in interval between voids, commonly the aim is to achieve an interval of three to four hours between voids and 3) positive reinforcement- - psychological support and encouragement is generally considered important and usually provided by health care professional . Frequency volume chart (FVC) records the time and volumes of voided for 24 hours by the women between the appointments. Four visits in 3 months with pelvic floor physical therapist, who is trained in the procedure, for educate and schedule voiding regimen.
  Interventions: Procedure: bladder training
- 3 (Active Comparator): The Pelvic floor muscle training (PFMT) protocol based on National Institute for health and clinical excellence (NICE clinical guideline 40, 2006), that the PFMT programs should comprise at least eight contractions performed three times per day, and the trial of supervised PFMT of at least 3 months' duration . Each appointment the women maid three sets of eight to 12 slow maximal contractions sustained for 6-8 second, and asked to made this protocol every day, and taught to contract these muscle to suppress urge filling. Four visits in 3 months with pelvic floor physical therapist, who is trained in the procedure, for reinforced pelvic floor muscles.
  Interventions: Procedure: pelvic floor muscle training
- 4 (Active Comparator): Four visits in 3 months with pelvic floor physical therapist, who is trained in the procedure, for pelvic floor muscle training and bladder training and lifestyle advice and information about good bladder and bowel habits.
  Interventions: Procedure: pelvic floor rehabilitation

INTERVENTIONS:
Procedure: tolterodine — Detrusitol SR 4 mg, 1 capsule for a day, 3 months.
  Arms: 1
Procedure: bladder training — Four visits in 3 months with pelvic floor physical therapist, who is trained in the procedure, for educate and schedule voiding regimen.
  Arms: 2
Procedure: pelvic floor muscle training — Four visits in 3 months with pelvic floor physical therapist, who is trained in the procedure, for reinforced pelvic floor muscles.
  Arms: 3
Procedure: pelvic floor rehabilitation — The Pelvic floor rehabilitation protocol based on bladder training protocol and PFMT and lifestyle advice and information about good bladder and bowel habits. Four visits in 3 months was made with pelvic floor physical therapist, who is trained in the procedure.
  Arms: 4

SUMMARY:
* Urinary Urge Incontinence (UUI) is the involuntary urine loss associated with a strong sensation to void.
* UUI usually associated with reduced bladder capacity.
* The pathophysiology is unclear.
* Pelvic floor muscle dysfunction and detrusor instability have been suggested as possible mechanisms.
* Standard treatment includes anticholinergic medication and behavior modification.
* The study aims to compare the long term effectiveness of 4 different approaches to the treatment of women with Urge Urinary Incontinence (UUI):

  1. Pelvic Floor Rehabilitation (includes muscle training+behavioral intervention+bladder training)
  2. Pelvic Floor muscle training alone
  3. Bladder Training alone
  4. Drug treatment with Tolterodine.
* Study variables will include: impairment ratings, quality of life, and cost-effectiveness.
* This study addresses three issues:

  1. The long term efficacy and cost-effectiveness of the various treatment options.
  2. To identify the factors involved in determining the effectiveness of drug or behavioral therapy.
  3. The pathophysiology of UUI. By subdividing the rehabilitation group into 3 arms, we hope to shed light on the mechanism of dysfunction. A better response in one group will help localize the problem to pelvic floor muscles or to detrusor instability.

DETAILED DESCRIPTION:
The study has 3 phases: Before treatment (phase I), immediately after 3 months of treatment (phase II), and 1 year post-entry (phase III)

Women with UUI will be divided randomly into one of the four treatment groups. Every subject will participate in 4 visits. The drug group treatment consists of administration of tolterodine SR 4 mg daily for 3 months. Subjects who assigned to the pelvic floor rehabilitation, pelvic floor muscle training, and bladder training groups will be treated via 4 visits to a physical therapist, who is trained in the procedures. The chief researcher (RK) will be blinded to the treatment groups and will perform the outcome measures in all phases.

Study variables will include impairment ratings, quality of life, and cost-effectiveness

ELIGIBILITY:
Inclusion Criteria:

* complaints of urinary leakage > 3 in last month (not stress incontinence)
* functionally independent subjects

Exclusion Criteria:

* urinary tract infection
* urogenital prolapse
* unstable diabetes
* neurological or psychiatric disease
* narrow angle glaucoma
* after colposuspension or sling surgery
* Mini Mental State Examination <24

Ages: 45 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2007-06; Primary Completion 2012-01 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Number of micturitions in a 24 hour bladder diary and number of urge urinary incontinence episodes by subjects' reports per week. | Phase I, II, and III

SECONDARY OUTCOMES:
cost-effectiveness | 1 year
Health service utilization | 1 year
underclothing pad use | Phase I, II, and III
change in physical activity and smoking | Phase I, II, and III
missed days at work | 1 year
Maximum voided volume, as obtained from 24 hours bladder diary | Phase I, II, III
side effects from list of 10 possible effects: dry mouth, constipation, side effects from list of 10 possible effects: dry mouth, constipation, sleepiness, fatigue, blurred vision, dizziness, urinary difficulty, tachycardia, headache and low back pain | Phase I, II, and III
quality of life measured by I-QoL | Phase I, II, and III
visual analogue scale (VAS) use in urogynecological research | Phase I, II, and III
Incontinence Severity Index (ISI) | Phase I, II, and III
functional status as measured by Late Life Function and Disability Instrument | Phase I, II, and III
Depression status as measured by Center for Epidemiological Studies Depression scale (CES-D) | Phase I, II, and III
Cost benefit | 1 year
Maximum voluntary contraction fo pelvic floor muscle, graded 1-5 by Oxford scale | Phase I, II, and III

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Kafri, MSc PT, Principal Investigator — Maccabi Healthcare Services, Israel
Locations (1):
- Rehabilitation and Physical Therapy Center, Maccabi Healthcare Services, Rishon LeZiyyon, Israel

REFERENCES:
- [Derived] Funada S, Yoshioka T, Luo Y, Sato A, Akamatsu S, Watanabe N. Bladder training for treating overactive bladder in adults. Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD013571. doi: 10.1002/14651858.CD013571.pub2. PMID 37811598